CLINICAL TRIAL: NCT05682105
Title: Detection of Jaundice From Ocular Images Via Deep Learning : a Prospective, Multicenter Cohort Study
Brief Title: Detection of Jaundice From Ocular Images Via Deep Learning
Status: Unknown | Type: Observational
Last Known Status: Active, not recruiting
Sponsor: Sun Yat-sen University (Other)
Collaborators: Third Affiliated Hospital, Sun Yat-Sen University (Other); Affiliated Huadu Hospital of Southern Medical University (Unknown); Aikang Health Care (Unknown)
Responsible Party: Principal Investigator, Haotian Lin, Principal Investigator, Sun Yat-sen University
Other Study IDs: AEHD-2022
Record Dates: First submitted 2022-12-26; First posted 2023-01-12 (Actual); Last update posted 2023-01-12 (Actual); Status verified 2023-01

CONDITIONS: Ophthalmology; Artificial Intelligence; Hepatobiliary Disease
Keywords: Ophthalmology; Artificial Intelligence; ocualr image; Jaundice
MeSH Terms: conditions — Digestive System Diseases; Jaundice

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Development dataset: Slit-lamp images collected from the Department of Hepatobiliary Surgery of the Third Affiliated Hospital of Sun Yat-sen University(HTH)， Affiliated Huadu Hospital of Southern Medical University(HDH)， and Nantian Medical Centre of Aikang Health Care (NMC).
- Testing dataset: Slit-lamp and smartphone images collected from the Department of Infectious Diseases, Third Affiliated Hospital of Sun Yat-sen University（ITH）， Huanshidong Medical Centre of Aikang Health Care， the Medical Centre of the Third Affiliated Hospital of Sun Yat-sen University(MCH).

SUMMARY:
Our study presents a detection model predicting a diagnosis of jaundice (clinical jaundice and occult jaundice) trained on prospective cohort data from slit-lamp photos and smartphone photos, demonstrating the model's validity and assisting clinical workers in identifying patient underlying hepatobiliary diseases.

DETAILED DESCRIPTION:
This study demonstrated that deep learning models could detect jaundice using ocular images in blood levels with reasonable accuracy, providing a non-invasive method for jaundice detection and recognition. This algorithm can assist clinical surgeons with daily follow-up visits and provide referral advice. It also highlights the algorithm's potential smartphone application in sizeable real-world population-based disease-detecting or telemedicine programs.

ELIGIBILITY:
Inclusion Criteria:

* The quality of slit-lamp images should be clinical acceptable. More than 90% of the slit-lamp image area, including three central regions (sclera, pupil, and lens) are easy to read and discriminate.

Exclusion Criteria:

* Images with light leakage (>10% of the area), spots from lens flares or stains, and overexposure were excluded from further analysis

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: This prospective, multicentre, observational study was led by Zhongshan Ophthalmic Centre (ZOC), Sun Yat-sen University, and conducted in three phases to collect data from participants from three surgery departments and three medical examination centres, including the Department of Hepatobiliary Surgery of the Third Affiliated Hospital of Sun Yat-sen University (HTH; Guangzhou, China), the Department of Infectious Diseases, Third Affiliated Hospital of Sun Yat-sen University (ITH; Guangzhou, China), the Department of Infectious Diseases, the Affiliated Huadu Hospital of Southern Medical University (HDH; Guangzhou, China), the Medical Centre of the Third Affiliated Hospital of Sun Yat-sen University(MCH; Guangzhou, China), Nantian Medical Centre of Aikang Health Care (NMC), and Huanshidong Medical Centre of Aikang Health Care (HMC).
Sampling Method: Probability Sample
Enrollment: 1633 (Actual)
Dates: Start 2018-12-01 (Actual); Primary Completion 2022-10-30 (Actual); Study Completion 2023-06-30 (Estimated)

PRIMARY OUTCOMES:
area under the receiver operating characteristic curve of the deep learning system | baseline
  The investigators will calculate the area under the receiver operating characteristic curve of deep learning system

SECONDARY OUTCOMES:
sensitivity and specificity of the deep learning system | baseline
  The investigators will calculate the sensitivity and specifity of deep learning system

CONTACTS AND LOCATIONS:
Locations (1):
- Zhongshan Ophthalmic Center, Guangzhou, Guangdong, China